CLINICAL TRIAL: NCT01958606
Title: High Intensity Interval Training in Chronic Stroke
Acronym: HIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: American Physical Therapy Association (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Brett Kissela, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIT in chronic stroke
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Exercise; Intensity; Gait
MeSH Terms: conditions — Stroke; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-intensity interval training (HIT) (Experimental): Treadmill exercise using bursts of concentrated effort alternated with recovery periods
  Interventions: Other: High-intensity interval training (HIT)
- Traditional aerobic training (Active Comparator): Moderate intensity continuous aerobic exercise on a treadmill
  Interventions: Other: Traditional Aerobic Training

INTERVENTIONS:
Other: High-intensity interval training (HIT) — Treadmill exercise using bursts of concentrated effort alternated with recovery periods
  Arms: High-intensity interval training (HIT)
Other: Traditional Aerobic Training — Moderate intensity continuous aerobic exercise on a treadmill
  Arms: Traditional aerobic training

SUMMARY:
The objective of this study was to compare the effectiveness of high intensity interval training (HIT) and traditional aerobic training for persons with stroke.

DETAILED DESCRIPTION:
Participants were randomized to either HIT or traditional aerobic training; each 25 minutes, 3 times per week for 4 weeks. Outcomes were measured before and after training by a blinded rater.

ELIGIBILITY:
Inclusion Criteria:

* 1) age 35-90 years
* 2) unilateral stroke experienced >6 months prior to enrollment
* 3) able to walk 10m overground with assistive devices as needed and no physical assistance
* 4) able to walk 3 minutes on the treadmill at >.13m/s (0.3mph) with no aerobic exercise contraindications
* 5) stable cardiovascular condition (American Heart Association class B, allowing for aerobic capacity <6 metabolic equivalents)
* 6) discharged from formal rehabilitation

Exclusion Criteria:

* 1) significant resting ECG abnormalities
* 2) evidence of significant arrhythmia or myocardial ischemia on treadmill ECG stress test
* 3) hospitalization for cardiac or pulmonary disease within 3 months
* 4) pacemaker or implanted defibrillator
* 5) lower extremity claudication
* 6) unable to communicate with investigators or correctly answer consent comprehension questions
* 7) severe lower extremity spasticity (Ashworth >2)
* 8) lower extremity weight bearing pain >4/10 on visual analogue scale

For the transcranial magnetic stimulation substudy, additional exclusions will also be applied. These include large cerebral infarcts or other structural defects with the potential to increase seizure risk, uncontrolled seizures, metal implants and previous craniotomy.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Kissela, MD, Principal Investigator — University of Cincinnati; Kari Dunning, PhD, PT, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Started | 13 | 5
Completed | 11 | 5
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9) | 57 (12) | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 7 | 2 | 9
Comfortable gait speed, m/s [Mean (Standard Deviation); unit: m/s] | 0.63 (0.48) | 0.76 (0.36) | 0.67 (0.44)
Peak oxygen consumption rate, ml/kg/min [Mean (Standard Deviation); unit: ml/kg/min] | 16.0 (4.0) | 21.6 (4.0) | 17.7 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Aerobic Capacity (VO2-peak)
Time Frame: Baseline and 4 weeks
Population: on treatment analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/kg/min
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 11 | 5
ml/kg/min | 2.2 [-0.05 to 4.5] | -1.3 [-4.7 to 2.1]

2. Secondary Outcome: Change in Submaximal Aerobic Capacity (VO2 at Ventilatory Threshold)
Time Frame: Baseline and 4 weeks
Population: ventilatory threshold was not identifiable for one participant
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/kg/min
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 10 | 5
ml/kg/min | 4.4 [3.1 to 5.7] | 0.6 [-1.3 to 2.5]

3. Secondary Outcome: Change in Gait Velocity (10 Meter Walk Test)
Time Frame: Baseline and 4 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: m/s
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 11 | 5
m/s | 0.10 [0.06 to 0.14] | 0.02 [-0.03 to 0.08]

4. Secondary Outcome: Change in 6-Minute Walk Test
Description: distance walked in 6 minutes
Time Frame: Baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 11 | 5
meters | 15 [1 to 29] | 15 [-6 to 36]

5. Secondary Outcome: Change in Gait Economy (Mean Oxygen Uptake at Comfortable Walking Speed)
Description: mean oxygen uptake at comfortable walking speed reported in units mLO2 per kilogram body weight per meter
Time Frame: Baseline and 4 weeks
Population: Subjects with available data
Measure: Mean (95% Confidence Interval); unit: mLO2/kg/m
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 9 | 5
mLO2/kg/m | -0.10 [-0.17 to -0.03] | -0.01 [-0.10 to 0.09]

6. Secondary Outcome: Change in Fastest Treadmill Speed (Steep Ramp Test)
Description: fastest safe treadmill walking speed
Time Frame: Baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: meters per second
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 11 | 5
meters per second | 0.36 [0.25 to 0.47] | 0.07 [-0.10 to 0.24]

7. Secondary Outcome: Change in Fractional Utilization
Description: Metabolic cost of gait as a percentage of aerobic capacity
Time Frame: Baseline and 4 weeks
Population: Subjects with available data
Measure: Mean (95% Confidence Interval); unit: percentage of aerobic capacity
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 8 | 5
percentage of aerobic capacity | -36.8 [-49.3 to -24.3] | -8.8 [-24.7 to -7.0]

8. Other Pre Specified Outcome: Change in Self-Efficacy and Outcome Expectations for Exercise Scale
Time Frame: Baseline and 4 weeks
Population: Outcome measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Change in Montreal Cognitive Assessment
Time Frame: Baseline and 4 weeks
Population: Measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: Change in Gait Kinematics/Kinetics From Baseline to 4 Weeks
Description: 3D motion capture and force plates
Time Frame: Baseline and 4 weeks
Population: Measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: Change in Gait Kinematics/Kinetics From Baseline to Post Session 1
Description: 3D motion capture and force plates
Time Frame: Baseline and after session 1
Population: measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Change in Gait Kinematics/Kinetics During Session 1
Description: 3D motion capture and force plates
Time Frame: During session 1
Population: measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Change in Transcranial Magnetic Stimulation (TMS) Responses From Baseline to 4 Weeks
Description: Primary variable is motor threshold (MT). Secondary variables include: motor evoked potential amplitude/latency, corticomotor map size and volume and intracortical inhibition
Time Frame: Baseline and 4 weeks
Population: measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: Change in Transcranial Magnetic Stimulation (TMS) Responses Associated With Training Session 2
Description: Primary variable is motor threshold (MT). Secondary variables include: motor evoked potential amplitude/latency and intracortical inhibition
Time Frame: Before and after training session 2
Population: measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Change in Transcranial Magnetic Stimulation (TMS) Responses Associated With Training Session 12
Description: as for outcome 14
Time Frame: Before and after training session 12
Population: measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: Change in Daily Physical Activity (Activity Monitor)
Time Frame: Baseline and 4 weeks
Population: measure not used
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: Change in Stroke Impact Scale
Description: Cognition Domain Score of Stroke Impact Scale. Scores range from 0 to 100 (higher is better) and represent a sum of scores from multiple questions related to cognition.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale from 0-100
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Number analyzed (Participants) | 11 | 5
units on a scale from 0-100 | 9.4 (15) | 0.7 (5.9)

ADVERSE EVENTS:
Arm/Group | High-intensity Interval Training (HIT) | Traditional Aerobic Training
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/5
Other Adverse Events (participants affected / at risk) | 9/13 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-intensity Interval Training (HIT) (N=13) | Traditional Aerobic Training (N=5)
Joint/muscle soreness (Musculoskeletal and connective tissue disorders) | 7 (10) | 2 (6)
Fatigue (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Light-headedness (Vascular disorders) | 2 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Other injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No